CLINICAL TRIAL: NCT06627595
Title: Impact of Physical Activity on Immunotherapy-induced Toxicities in Melanoma Management
Acronym: APiTOXMM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0195
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Melanoma; Immunotoxicity
Keywords: physical activity; melanoma; immunotherapy; anti-PD-1; anti-CTLA4; immunotoxicity
MeSH Terms: conditions — Melanoma; Motor Activity | interventions — Immunotherapy; pembrolizumab; Nivolumab; Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with no physical activity / low physical activity: Patients with low score according to the IPAQ questionnaire at baseline. This is the lowest level of physical activity.
  Interventions: Drug: Immunotherapy
- Patients with moderate to high physical activity: Patients with moderate or high score according to the IPAQ questionnaire at baseline.
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Patients will be treated in accordance with the guidelines for melanoma treatment.
  Other Names: pembrolizumab; nivolumab; ipilimumab

SUMMARY:
Management of melanoma is based on primary excision of the tumor. In cases of melanoma with poor prognosis criteria, or when it is locally advanced or metastatic, there is an indication for the implementation of adjuvant therapy, which may, in this context, be immunotherapy.

Immunotherapies are treatments that have revolutionized the prognosis of patients with melanoma. These are therapies that work by stimulating the immune system to enhance the anti-tumor response. Their toxicities are represented by immune-mediated toxicities, similar to true autoimmune diseases.

Adapted physical activity as supportive care in oncology is expanding. From a pathophysiological perspective, physical activity is thought to modulate the immune system (by reducing inflammation, restoring immune surveillance, stimulating anti-tumor responses through the induction of T cell proliferation, modulating the gut microbiota, and influencing tumor microenvironment cells, etc.).

The modulation of the immune system by physical activity may also allow us to hypothesize a modulation of the toxicities induced by immune checkpoint inhibitors. We wish to study this hypothesis in patients with advanced melanoma who are candidates for immunotherapy.

Originality and Innovative Aspects:

Physical activity as supportive care in oncology has developed significantly in recent years. However, adapted physical activity (APA) is currently only offered at one center in France (CHU de Lille).

In addition to the probable impact on patients' quality of life, if we find evidence supporting a reduction in treatment-related toxicities for melanoma through physical activity, it would be even more interesting to introduce APA at the CHU of Montpellier.

Primary and Secondary Objectives:

Primary Objective: To analyze the association between the level of physical activity (estimated by the IPAQ questionnaire) at the initiation of immunotherapy and the occurrence of adverse effects at 6 months after starting treatment in adult patients with melanoma.

Secondary Objectives:

Analyze the association between physical activity level and treatment efficacy of immunotherapy in adult melanoma patients.

Describe the quarterly evolution of patients' general condition through measurement of WHO status and BMI.

Assess the evolution of patients' general condition: WHO status and BMI at treatment introduction, after 3 months, and at 6 months of treatment.

Study the evolution of patients' quality of life during their treatment based on their physical activity level, using the QLQ-C30 questionnaire.

Preliminary study:

We aim to evaluate the correlation between self-reported physical activity by patients and their actual physical activity. To obtain an objective measurement of patients' physical activity level, we plan to work with the CARTIGEN platform and offer a small number of included patients (maximum of 50) to wear wrist actimeters for one week before treatment initiation. We will then analyze these data to determine patients' baseline physical activity levels and compare them with the data collected via questionnaires.

This is a prospective cohort study within the context of analytical epidemiological research. It is a bicentric study: CHRU Montpellier - Saint-Eloi Hospital and ICM Val d'Aurelle.

Using the collected data on patients' physical activity levels (IPAQ questionnaire), we will compare two groups: patients who experienced immuno-toxicities without physical activity versus those with moderate or high physical activity.

We will also analyze treatment efficacy in these two groups, patients' quality of life, and the evolution of their general condition.

Procedure:

Inclusion is planned at day 0 (D0), with physical activity (IPAQ3) and quality of life (QLQ-C30) questionnaires, along with clinical and oncological evaluation.

A follow-up visit at month 3 (M3) will include reassessment of clinical and oncological status, followed by another visit at month 6 (M6) for further clinical, oncological, physical activity, and quality of life reassessment.

The inclusion period is expected to last 18 months.

Outcomes / Perspectives:

If we consider that physical exercise may help mitigate the toxic effects of treatments-an aspect we wish to explore through this project-it would be relevant to introduce adapted physical activity (APA) sessions supervised by a specialized instructor within the Dermatology Day Hospital at the CHU of Montpellier.

Implementing APA in the context of onco-dermatology will strengthen the multidisciplinary approach of the CHU.

Collaboration between healthcare professionals, including specialized APA instructors, will foster effective care coordination.

This initiative is part of a holistic approach to patient care, integrating complementary interventions to address physical, psychological, and social needs.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* ECOG performance status inferior or equal to 3
* patient with a melanoma confirmed histologically/pathologically
* indication for initiating treatment with anti-PD1 immunotherapy or anti-PD1 + anti-CTLA4

Exclusion Criteria:

* patient unable to read and/or write
* inability to follow up with the patient during the study period
* refusal to participate after a reflection period
* medical contraindication to initiating immunotherapy (active autoimmune disease requiring systemic treatment in the past 2 years, active infection, etc.)
* not affiliated with a social security system
* patient under legal protection, guardianship, or curatorship
* person participating in another study that includes an ongoing exclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18 years or older, newly diagnosed with melanoma with an indication for treatment initiation by immunotherapy (anti-PD1 or anti-PD1 + anti-CTLA4), in an adjuvant or metastatic setting. Only incident cases will be included. Patients treated at Montpellier University Hospital (CHU) or the Montpellier Cancer Institute (ICM)
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Immunotoxicity | From the time of enrollment until 6 months following the initiation of treatment
  Occurrence of immune-induced side effects

SECONDARY OUTCOMES:
Efficacy of immunotherapy | From the time of enrollment until 6 months following the initiation of treatment
  Tumoral response to immunotherapy

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - Institut du Cancer de Montpellier (ICM), Montpellier

IPD SHARING:
Plan to Share IPD: No